CLINICAL TRIAL: NCT01476293
Title: Non-invasive Optical Medical Device for Monitoring and Detecting Peripheral Intravenous Infusion Sites for Infiltration and Extravasation in Subjects Receiving Continuous Fluids
Brief Title: Monitoring the Peripheral Intravenous Infusion Site for Infiltration and Extravasation
Status: Completed | Type: Observational
Sponsor: ivWatch, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: ivWatch-CT-001
Record Dates: First submitted 2011-11-09; First posted 2011-11-22 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2011-11

CONDITIONS: Infiltration; Extravasation; IV Infiltration; IV Extravasation; Extravasation of Diagnostic and Therapeutic Materials
Keywords: Infiltration; Extravasation; Leaking; PIV Infiltration; IV Infiltration; Optical Detection of Infiltration; Optical Monitoring
MeSH Terms: conditions — Extravasation of Diagnostic and Therapeutic Materials

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study to to monitor the peripheral intravenous (PIV) site on subjects receiving continuous IV fluids for infiltration and extravasation events. Infiltration is an indication that the PIV is leaking fluids outside of the vascular system. The study hypothesis is to demonstrate that changes in the optical signals of the non-invasive monitoring medical device will detect infiltration and extravasation events.

ELIGIBILITY:
Inclusion Criteria:

* signed consent
* patient age under 12
* PIV with continuous fluids

Exclusion Criteria:

* no consent
* patient age over 12
* PIV fluids not continuous

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects will be recruited from Cincinnati Children's Hospital Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Test performance of optical device for monitoring intravenous infusion site for infiltration. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Doellman, RN, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Sylvia Rineair, MSHA, BSN, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Neil Johnson, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Michael Spigarelli, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States